CLINICAL TRIAL: NCT05767879
Title: Open Label Phase 2 Study Neo-Adjuvant BRAF/MEK Inhibition Followed by Surgery and Adjuvant BRAF/MEK Inhibition in In-transit Melanoma Metastases (NASAM)
Brief Title: (Neo)Adjuvant BRAF/MEK Inhibition in pN1c Melanoma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Leiden University Medical Center (Other)
Collaborators: Pierre Fabre Laboratories (Industry)
Responsible Party: Principal Investigator, HW Kapiteijn, Phd, Leiden University Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NL77905.058.21; 2021-002285-40 (EudraCT Number)
Record Dates: First submitted 2022-08-16; First posted 2023-03-14 (Actual); Last update posted 2023-03-14 (Actual); Status verified 2023-03

CONDITIONS: Melanoma Stage III; In-Transit Metastasis of Cutaneous Melanoma
Keywords: Targeted therapy; In-transit; Melanoma; Neo-adjuvant
MeSH Terms: conditions — Melanoma | interventions — encorafenib; binimetinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Neo adjuvant BRAF/MEK inhibition in pN1c Melanoma (Experimental): Neo adjuvant BRAF/MEK inhibition (encorafenib/binimetinib).
  Patients receive encorafenib 450 mg once daily for a period of 8 weeks. Patients receive 45 mg binimetinib twice daily for a period of 8 weeks. After the neo-adjuvant therapie, patients will receive encorafenib 450 mg once daily fand binimetinib 45mg twice daily for 44 weeks.
  Interventions: Drug: Encorafenib + Binimetinib

INTERVENTIONS:
Drug: Encorafenib + Binimetinib — In the open label phase II study, the combination of BRAF/MEK inhibition with encorafenib/binimetinib in the neo-adjuvant setting will be investigated.
  Furthermore, efficacy of adjuvant BRAF/MEK inhibition with encorafenib/binimetinib, for 44 weeks will be evaluated.

SUMMARY:
Phase 2 open-label single arm intervention study administering encorafenib/binimetinib in neo-adjuvant setting followed by surgery and subsequent adjuvant encorafenib/binimetinib in in-transit melanoma patients without lymph node and distant metastases.

DETAILED DESCRIPTION:
Phase 2 open-label single arm intervention study administering encorafenib/binimetinib in neo-adjuvant setting followed by surgery and subsequent adjuvant encorafenib/binimetinib in patients diagnosed solely with in-transit metastatic melanoma.

Primary objective is to determine the efficacy of neo-adjuvant encorafenib/binimetinib as measured by pathological response rate (partial-, complete- and no response). In the biopsy at week 0 the viability will be judged and will be graded according to the amount of tumor necrosis: >50% tumor necrosis with <50% viable tumor cells, <50% necrosis with >50% viable tumor cells and 100% necrosis without viable tumor cells. Partial response is defined as a decrease of at least 50% of the viable tumor cells and complete response as 100% decrease of tumor cells, whereas no response is defined as more than 50% of viable tumor cells present.

Secondary objectives are to assess efficacy of adjuvant BRAF/MEK inhibition, measured as local recurrence free survival (LRFS), distant metastases-free survival (DFMS), recurrence free survival (local and/or distant recurrence, RFS) and overall survival (OS). Additionally, the toxicity of the administered regimen will be assessed by analyzing the frequency- and type of adverse events, and occurrences of therapy interruption, dose reduction and or therapy cessation. Moreover, an exploration of drug measurements and ctDNA in blood and additional research of biopsies / resections will be done.

ELIGIBILITY:
Inclusion Criteria:

* Age over 18 years old
* World Health Organization (WHO) Performance Status 0 or I
* Primary cutaneous melanoma or unknown primary melanoma with pathologically confirmed in-transit metastatic melanoma
* Patients must have undergone complete disease staging including: PET-CT scan and MRI scan
* Patients must be medically fit to undergo surgery
* Patients must be able to take oral medication
* No prior anticancer systemic treatment (including chemotherapy, immunotherapy, oncolytic viral therapy, other systemic therapies)
* No prior radiotherapy to site of interest (surgical therapy is allowed; in order to obtain pathological information of the melanoma)
* Screening laboratory values must meet the following criteria: WBC ≥ 2.0x109/L, Neutrophils ≥ 1.0x109/L, Platelets ≥ 100 x109/L, Hemoglobin ≥ 6.5 mmol/L, AST ≤ 2.5 x ULN, ALT ≤ 2.5 x ULN, Total bilirubin ≤ 1.5 X ULN, INR and PTT in normal range, LDH < 2xULN. Serum creatinine ≤ 1.5 × ULN; or calculated creatinine clearance ≥ 50 mL/min by Cockcroft-Gault formula; or estimated glomerular filtration rate > 50 mL/min/1.73m2.
* Absence of additional severe and/or uncontrolled concurrent disease

Exclusion Criteria:

* Presence of regional lymph node metastases
* Presence of distant metastases
* Current treatment with antiretroviral drugs, herbal remedies and drugs that are strong inhibitors or inducers of CYP3A and CYP2C8
* Patients with active bacterial infections with systemic manifestations (malaise, fever, leukocytosis) are not eligible until completion of appropriate therapy
* Underlying medical conditions that, in the Investigator's opinion, will make the administration of study treatment hazardous or obscure the interpretation of toxicity determination or adverse events
* History of congestive heart failure, active cardiac conditions, including unstable coronary syndromes (unstable or severe angina, recent myocardial infarction), significant arrhythmias and severe valvular disease must be evaluated for risks of undergoing general anesthesia. Furthermore, enlarged QTc interval, uncontrolled hypertension, poor left ventricular function (< 50%, as determined by MUGA scan) and recent thromboembolic or cerebral event.
* History of central serous retinopathy or retinal vein occlusion
* Active intestinal disease interfering with oral drug absorption
* Patients who are unable to be temporally removed from chronic anti-coagulation therapy for operation
* (Neo)Adjuvant BRAF/MEKi for pN1c melanoma, version 5, 31 October 2021
* Other malignancy within 2 years prior to entry into the study, except for treated non-melanoma skin cancer and in situ cervical carcinoma
* Patient must not have active hepatitis B, and/or active hepatitis C infection given concerns for drug interactions or increased toxicities. Testing is not required
* Patient must not have any known history of acute or chronic pancreatitis
* Patient must not have any concurrent neuromuscular disorder that is associated with elevated creatine kinase (CK) (e.g., inflammatory myopathies, muscular dystrophy, amyotrophic lateral sclerosis, spinal muscular atrophy
* Pregnancy or nursing

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Estimated)
Dates: Start 2022-01-01 (Actual); Primary Completion 2026-01-01 (Estimated); Study Completion 2026-01-01 (Estimated)

PRIMARY OUTCOMES:
Efficacy of neo-adjuvant encorafenib/binimetinib | 8 weeks
  Primary outcome is to determine the efficacy of neo-adjuvant eEncorafenib/bBinimetinib as measured by pathological response rate (partial-, complete- and no response). In the biopsy at week 0 the viability will be judged and will be graded according to the amount of tumor necrosis: >50% tumor necrosis with <50% viable tumor cells, <50% necrosis with >50% viable tumor cells and 100% necrosis without viable tumor cells. Partial response is defined as a decrease of at least 50% of the viable tumor cells, and complete response is defined as more than 90% a decrease of more than 90% of the tumor cells, whereas no response is defined as more than 50% of viable tumor cells present.

SECONDARY OUTCOMES:
Evaluate efficacy of treatment related toxicity | 52 weeks
  analyzing the frequency- and type of adverse events, and occurrences of therapy interruption, dose reduction and or therapycessation. Adverse events severity will be graded according to the National Cancer Institute's Common Terminology Criteria for Adverse Events, version 5.0. Adverse events associated with BRAF/MEK inhibition will be termed as treatment related or potentially treatment related, adverse events which are not known class effects of BRAF/MEK inhibitors will be described as adverse events not treatment related. Adverse event assessment will take place from therapy initiation up to completion of adjuvant treatment (week 44) and 30 das after.
Efficacy of adjuvant encorafenib/binimetinib - local recurrece free survival (LRFS) | 44 weeks
  To assess efficacy of adjuvant BRAF/MEK inhibition by analyzing the surgical site clinically (bimonthly) and radiologically (every 4 months) during the adjuvant treatment.
  Local disease recurrence is defined as pathologically confirmed metastasic melanoma in scar tissue and or recurrence of melanoma within 2cm of the surgical scar of primary melanoma of the previously removed melanoma.
  Local disease recurrence will be measured from start of adjuvant therapy up to disease recurrence confirmation.
Efficacy of adjuvant encorafeninb/binimetinib - distant metastases-free survival (DFMS) | 44 weeks
  To assess efficacy of adjuvant BRAF/MEK inhibition by analyzing the surgical site clinically (bimonthly) and radiologically (every 4 months) during the adjuvant treatment.
  Distant metastases free survival (DFMS) is defined as the moment of pathologically and or radiologically disease confirmation.
  Distant metastatic disease includes, distant lymph nodes and organs. Distant metastatic free survival will be calculated using the start of therapy up to the moment of distant metastatic disease confirmation or last follow-up moment.
Efficacy of adjuvant encorafeninb/binimetinib - overall survival | 44 weeks
  To assess efficacy of adjuvant BRAF/MEK inhibition by analyzing the surgical site clinically (bimonthly) and radiologically (every 4 months) during the adjuvant treatment.
  Overall survival is defined as the moment of primary melanoma up to decease.
Efficacy of adjuvant encorafeninb/binimetinib - treatment related survival | 44 weeks
  To assess efficacy of adjuvant BRAF/MEK inhibition by analyzing the surgical site clinically (bimonthly) and radiologically (every 4 months) during the adjuvant treatment.
  The moment of start of adjuvant therapy up to decease or last follow-up moment.

CONTACTS AND LOCATIONS:
Locations (1):
- Leiden University Medical Center, Leiden, South Holland, Netherlands

IPD SHARING:
Plan to Share IPD: No